CLINICAL TRIAL: NCT03241784
Title: Expansion and Infusion of T-Regulatory Cells in Amyotrophic Lateral Sclerosis
Brief Title: T-Regulatory Cells in Amyotrophic Lateral Sclerosis
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Stanley H. Appel, MD (Other)
Responsible Party: Sponsor-Investigator, Stanley H. Appel, MD, TMHPO Chairman & Principal Investigator, The Methodist Hospital Research Institute
Organization: The Methodist Hospital Research Institute (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00013616
Record Dates: First submitted 2017-07-27; First posted 2017-08-07 (Actual); Last update posted 2018-03-26 (Actual); Status verified 2018-03

CONDITIONS: ALS (Amyotrophic Lateral Sclerosis)
Keywords: ALS; T-Regulatory Cells
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — Interleukin-2

STUDY DESIGN:
Intervention Model Description: Autologous infusion of expanded T-regulatory lymphocytes during early and late phases of ALS disease in patients with varying rates of disease progression.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment arm (Experimental): All subjects are enrolled in the one arm consisting of infusions of autologous T-regulatory lymphocytes at a dose of 1x10 to the sixth/kg and subcutaneous injections of Interleukin-2 at a dose of 2x10 to the fifth IU/m2 three times a week.
  Interventions: Biological: Autologous T-regulatory lymphocytes; Biological: Interleukin-2

INTERVENTIONS:
Biological: Autologous T-regulatory lymphocytes — intravenous administration of Autologous T-regulatory lymphocytes at a dose of 1x10 to the sixth /kg.
Biological: Interleukin-2 — Subcutaneous Interleukin-2 at a dose of 2x10 to the fifth IU/m2, three times a week.
  Other Names: IL-2

SUMMARY:
This is an open-label pilot study to determine the safety and tolerability of infusions of autologous CD4+ CD25+ regulatory T cells with concomitant subcutaneous IL-2 injections in 4 subjects with ALS.

DETAILED DESCRIPTION:
This Pilot Study will consist of 4 ALS subjects who will undergo 4 infusions of autologous expanded Tregs with concomitant subcutaneous injections of IL-2 (2 x 105 IU/m2) 3 times weekly for 52 weeks or at least until such time that interim analyses can confirm or negate its benefit.

During the enrollment period up to four subjects will be recruited from patients known to our clinic for screening, baseline measures and leukapheresis. The Treg cell manufacturing will be performed in a GMP laboratory. The first subject will receive infusions of their expanded Tregs (1x106 /kg) with concomitant subcutaneous IL-2 injections (2 x 105 IU/m2) 25 days (+/- 2 days) post leukapheresis. The 2nd subject will begin after the first subject has completed the first 4 weeks and has experienced no untoward effects during this period. Once subjects #1 and #2 have completed the first 4 weeks and no toxic events have occurred they will therefore be considered safely past the first milestone and subject #3 will begin infusions. After subject #3 has completed the first 4 weeks with no untoward effects, subject #4 may begin infusions with the below modified schedule:

The 4th subject will undergo infusion of autologous expanded Tregs once every four weeks (+/- 2 days) for a total of four infusions, with concomitant subcutaneous injections of IL-2 (2 x 105 IU/m2) 3 times weekly. In addition, subject #4 will begin subcutaneous IL-2 injections 4 weeks before his first autologous Treg infusion. An additional office visit will take place 2 weeks after initiating IL-2 for clinical evaluation, scoring and blood draw. Office visits will then be completed every two weeks while the subject is receiving Treg infusions for clinical evaluation, scoring, and blood draws. Then, the subject will be seen in office visits once per month for one year total for clinical evaluation, scoring, and blood draws.

In addition, subjects #1, 2 and 3 will repeat the leukapheresis (under a separate protocol) and undergo Treg infusions at the modified schedule of every 4 weeks, with concomitant subcutaneous injections of IL-2 (2 x 105 IU/m2) 3 times weekly. The subjects will be called on Day 7, and 21. Office visits will be completed on the day after infusions and every two weeks while the subjects are undergoing Treg infusions for clinical evaluation, scoring, and blood draws. The subjects will then be seen during office visits once per month for one year total from their initial baseline visit for clinical evaluation, scoring, and blood draws

Monthly interim analyses will monitor the subjects using validated ALS scales such as the ALSFRS-R and Appel Scale, which incorporates muscle strength and dysfunction, activities of daily living and pulmonary function. The analyses will also include interim medical history and physical exam, EKG when indicated, safety labs (such as CBC, chemistry, liver function, T4 and TSH) as well as more technical research labs such as T Regulatory Cell, Th1 and Th17 counts, FoxP3 RNA expression, and Treg Suppression Assays. A PT/PTT will be performed only if the subject has an abnormal coagulation result at baseline or if the subject is on anti-coagulation therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older.
2. Sporadic or familial ALS diagnosed as possible, laboratory-supported probable, probable, or definite as defined by revised El Escorial criteria (Appendix 1).
3. Subjects must not have taken riluzole for at least 30 days, or be on a stable dose of riluzole for at least 30 days (riluzole-naïve subjects are permitted in the study).
4. Capable of providing informed consent and following trial procedures.
5. Geographically accessible to the site.
6. Women must not be able to become pregnant (e.g. post-menopausal, surgically sterile, or using adequate birth control methods) for the duration of the study and three months after study completion. Adequate contraception includes: abstinence, hormonal contraception (oral contraception, implanted contraception, injected contraception or other hormonal (patch or contraceptive ring, for example) contraception), intrauterine device (IUD) in place for ≥ 3 months, barrier method in conjunction with spermicide, or another adequate method.
7. Subjects must agree not to take live attenuated vaccines (including seasonal flu vaccine) 30 days before blood collection.
8. Available autologous Tregs product with greater than or equal to 50% expression of CD4, CD25 and FoxP3 determined by flow-cytometry.
9. Subjects must have been previously evaluated and followed clinically by a neuromuscular specialist at Houston Methodist Neurological Institute
10. Normal Alanine aminotransferase level (ALT)
11. Normal Serum creatinine level

Exclusion Criteria:

1. Prior use of cells therapies
2. Concurrent use of other experimental ALS therapies
3. Pregnant or breastfeeding or planning to become pregnant or planning a partner's pregnancy.
4. Other unstable medical or psychiatric illness
5. Known immune deficiency or history of lymphoma or leukemia
6. History of lymphopenia.
7. History of acquired or inherited immune deficiency syndrome, including leukopenia.
8. History of severe untreated chronic obstructive sleep apnea.
9. FVC less than 50% predicted at screening.
10. Exposure to any other agent currently under investigation for the treatment of subjects with ALS (off-label use or investigational) within 30 days of the Baseline Visit.
11. The presence of unstable psychiatric disease, cognitive impairment, or dementia that would impair ability of the subject to provide informed consent, according to the PI's judgment, or a history of active substance abuse within the prior year.
12. Clinically significant history of cardiac, oncologic, hepatic, or renal dysfunction, or other medically significant illness.
13. The presence of any immunologic or autoimmune disease
14. Severe cardiac dysfunction defined clinically, or as a left ventricular ejection fraction less than 40% of predicted or abnormal EKG findings.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Estimated)
Dates: Start 2016-05-16 (Actual); Primary Completion 2018-02 (Actual); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | Baseline to two years
  Clinical laboratory blood tests are standard to assure safety in clinical trials. Complete blood count, chemistry, liver function, throxine (T4) and thyroid stimulating hormone (TSH) will be assessed for normal reference ranges and abnormal (not clinically significant) results. Clinically abnormal results will be documented as adverse events as per CTCAE v4.0.

SECONDARY OUTCOMES:
AALS (Appel ALS) Scale | Baseline to week 15
  The AALS is a published, validated instrument that consists of five sub-scores: bulbar, respiratory, muscle strength, and lower extremity and upper extremity function. Each group is composed of individual tests. The total Appel ALS score is 30 for healthy subjects and 164 for those with maximum impairment. The rate of change in the Appel ALS Rating Scale is a significant predictor of survival for subjects with ALS.
ALSFRS-R (ALS Functional Rating Scale-Revised) | Baseline to week 15
  The ALSFRS-r (ALS Functional Rating Scale-revised) is an orally administered validated instrument using an ordinal rating scale used to determine the subject's assessment of their capability and independence in 12 functional activities. The scale addresses fine motor, gross motor, bulbar and respiratory function. The ALSFRS-r is used as a clinical assessment in ALS standard of care and in most ALS clinical trials.
T-Regulatory Cells | Baseline to 3 months post treatment for a total of two years from baseline
  Treg percentage (CD4+CD25+FOXP3+ cells) within the total CD4+ population will be assessed by multicolor flow cytometry.
Treg Suppression | Baseline to 3 months post treatment for a total of two years from baseline
  Treg suppressive function of T-effector (Teff) cells will be assessed by [3H]-thymidine incorporation. Correlation between changes in the rate of disease progression and the Treg percentage and function will be determined by Spearman's correlation analysis.
TH17 and Th1 lymphocytes | Baseline to 3 months post-treatment for a total of two years from baseline
  The percentage of Tregs, Th1 lymphocytes and Th17 lymphocytes will be assessed by multicolor flow cytometry.

OTHER OUTCOMES:
Pulmonary FVC - Exploratory Measure | Baseline to 3 months post-treatment for a total of two years from baseline
  FVC (Forced Vital Capacity). Reduction of pulmonary function is the primary source of morbidity and mortality in ALS. FVC testing will be used to monitor respiratory function. FVC measures the amount of air which can be forcibly exhaled from the lungs after taking the deepest breath possible.
Pulmonary MIP - Exploratory Measure | Baseline to 3 months post-treatment for a total of two years from baseline
  MIP (Maximum Inspiratory Pressure. Reduction of pulmonary function is the primary source of morbidity and mortality in ALS. MIP testing will be used to monitor respiratory function. MIP measures inspiratory muscle strength.
Tracheostomy- Exploratory Measure | Baseline to 3 months post-treatment for a total of two years from baseline
  Duration of tracheostomy-free survival

CONTACTS AND LOCATIONS:
Overall Officials: Stanley H Appel, MD, Principal Investigator — Houston Methodist Neurological Institute
Locations (1):
- Methodist Neurological Institute, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No